CLINICAL TRIAL: NCT06164301
Title: the Value of Early Post-operative Elemental Amino Acids in Critically Ill Obstetrics, and Its Contribution to the Concept of ERAS
Brief Title: Value of Early Post Operative Amino Acids in Critically Ill Obstetrics on Recovery Enhancement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FMASU R290/2023
Record Dates: First submitted 2023-11-21; First posted 2023-12-11 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-12

CONDITIONS: Malnutrition in Pregnancy; Malnutrition; Protein; Postpartum Disorder; Patient Satisfaction; Critical Illness
Keywords: critical illness; nutrition therapy; Enhanced Recovery After Surgery; Enhanced Recovery After Caesarean section
MeSH Terms: conditions — Kwashiorkor; Puerperal Disorders; Patient Satisfaction; Critical Illness

STUDY DESIGN:
Intervention Model Description: Patients will be assigned into either; A)Elemental Amino group ; post-operative within the first 3 hours the patient will receive 250 ml of elemental protein( 250 ml Peptamen = 6 scoops (55g) + 210ml water ) repeated at ( 6, 8 , 10 , 12 hours postoperative ) , Second day ordinary food will be supplemented by half the dose of the first day from elemental protein (250 ml / 6 hours ) or to the dose to achieve the daily protein adequacy 1.3 mg/kg/day. B) The standard group will be NPO till the return of bowel functions.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Elemental Amino group (Experimental): Elemental Amino group ; post-operative within the first 3 hours the patient will receive 250 ml of elemental protein( 250 ml Peptamen = 6 scoops (55g) + 210ml water ) repeated at ( 6, 8 , 10 , 12 hours postoperative ) in order to reach total protein in order to reach total protein 50 mg in the first 12 hour post-operative, Second day ordinary food will be introduced supplemented by half the dose of the first day from elemental protein (250 ml / 6 hours ) or to the dose to achieve the daily protein adequacy 1.3 mg/kg/day.
  Interventions: Dietary Supplement: Elemental amino-acids
- standard (Active Comparator): Standard group; The patients in this group will receive the standard protocol in which they will be made NPO till the return of bowel functions. Thereafter, water and clear fluids will be given followed by soft food and, eventually a regular diet.
  Interventions: Dietary Supplement: Elemental amino-acids

INTERVENTIONS:
Dietary Supplement: Elemental amino-acids — mono peptide oral protein formula

SUMMARY:
This is the first trial to assess the early elemental postoperative amino-acid load to meet the protein requirements in the first and second day postoperative to enhance the recovery of critically ill parturient (value on ERAS of critically ill obstetrics)

DETAILED DESCRIPTION:
The objective is to measure the effect of elemental amino acids in early post-operative period on reaching protein adequacy as well as energy intakes, gut function, clinical outcomes, and the quality of recovery.

All candidates will be assessed thoroughly by history and examination, and informed consent will be taken. All patients will be admitted to the obstetrics ICU. where degree of severity of the condition will be assessed and the relevant protocol of treatment will be started. All patients will receive the treatment algorithm of critically ill as follow; Prophylactic anticoagulation (Enoxaparin 40 mg once daily) when appropriate after surgeon consultation. Antibiotic as policy, Proton pump inhibitors (omeprazole 40 mg once daily), Other supportive medication according to the needs of the condition, For postoperative pain routine care in the form of use of paracetamol (10mg/kg/8 hrs), and non-steroidal anti-inflammatory(ketorolac 30 mg /12 hrs ) medication and nalbuphine will be used till comfort of the patient. All doses will be adjusted according to body weight and organ function when required. Base line laboratory indices will be withdrawn including; CBC, Metabolic profile, liver function profile, renal function profile, ABG, INR.

The eligible patients will be randomly assigned into one of two groups through the random numbers, the random numbers will be used by a pharmacist who will prepare the different regimen. the data collector will be blind about the grouping intervention. A)Elemental Amino group ; post-operative within the first 3 hours the patient will receive 250 ml of elemental protein( 250 ml Peptamen = 6 scoops (55g) + 210ml water ) repeated at ( 6, 8 , 10 , 12 hours postoperative ) in order to reach total protein in order to reach total protein 50 mg in the first 12 hour post-operative, Second day ordinary food will be introduced supplemented by half the dose of the first day from elemental protein (250 ml / 6 hours ) or to the dose to achieve the daily protein adequacy 1.3 mg/kg/day. B) Standard group; The patients in this group will receive the standard protocol in which they will be made NPO till the return of bowel functions. Thereafter, water and clear fluids will be given followed by soft food and, eventually a regular diet. Protein requirement in postpartum around 1g/kg reaching up to 1.9 gm/kg 11. The investigator will standardize the intake to 1.3g/kg.

In both groups intravenous fluid will be given according to hemodynamic in the form of ringer acetate with basal infusion 40ml/hr and will be adjusted according to hemodynamic parameters. In both groups, daily food and fluid record will be assessed by research assistant who will follow both the patient recall and the nurse record. The research assistant will be provided by written details in how to calculate protein and energy intake.

ELIGIBILITY:
Inclusion Criteria:

* Critically ill Female patients with cesarean section with or without hysterectomy that requires ICU admission pre or postoperative

Exclusion Criteria:

* Decompensated heart failure,
* Known allergy
* Tryptophan intolerance
* known inborn errors of metabolism of proteins as alkaptonuria
* severe hepatic dysfunction (failure)
* severe renal dysfunction (failure)
* severe coagulopathy or DIC
* circulatory shock or hemodynamic instability
* Lactose intolerance
* G6PD deficiency

Ages: 16 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Gender Based: Yes — pregnant female for cesarean section
Enrollment: 83 (Actual)
Dates: Start 2024-04-14 (Actual); Primary Completion 2025-12-20 (Actual); Study Completion 2026-01-20 (Actual)

PRIMARY OUTCOMES:
the protein intake | 24 hours postoperative. If the patient stay extended more than a day, the intake of second 24 hours will be calculated,
  total protein intake/day measurement tool is calculation based on protein content in the food intake list , and measured by gram/kg/day
The energy intake | 24 hours postoperative. If the patient stay extended more than a day, the intake of second 24 hours will be calculated
  total energy intake/day, The measurement tool is calculated by an experienced clinical nutrition pharmacist based on food and supplements intake in nursing records and patient recall, and measured by kcal/kg/day

SECONDARY OUTCOMES:
satisfaction and Patient reported outcome measures (PROMs) regarding recovery aspects (physical comfort- emotional state, physical independence and pain | After 48 hours or at discharge from ICU which comes first
  will be assessed using the Obstetric Quality of Recovery-10A survey tool and measured by units on the scale, it is 10 questions with answers on a scale from 0 to 10 where 0 =very poor and 10 = excellent. with cumulative score where <71= poor, 71-88= moderate, >88= excellent.

CONTACTS AND LOCATIONS:
Overall Officials: wessam selima, MD, Principal Investigator — assistant professor (lecturer)- Ain shams university
Locations (1):
- Ain shams university, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared on reasonable request

REFERENCES:
- [Background] Macones GA, Caughey AB, Wood SL, Wrench IJ, Huang J, Norman M, Pettersson K, Fawcett WJ, Shalabi MM, Metcalfe A, Gramlich L, Nelson G, Wilson RD. Guidelines for postoperative care in cesarean delivery: Enhanced Recovery After Surgery (ERAS) Society recommendations (part 3). Am J Obstet Gynecol. 2019 Sep;221(3):247.e1-247.e9. doi: 10.1016/j.ajog.2019.04.012. Epub 2019 Apr 14. PMID 30995461
- [Background] Looijaard WGPM, Denneman N, Broens B, Girbes ARJ, Weijs PJM, Oudemans-van Straaten HM. Achieving protein targets without energy overfeeding in critically ill patients: A prospective feasibility study. Clin Nutr. 2019 Dec;38(6):2623-2631. doi: 10.1016/j.clnu.2018.11.012. Epub 2018 Dec 17. PMID 30595377
- [Background] Meyer R, Foong RX, Thapar N, Kritas S, Shah N. Systematic review of the impact of feed protein type and degree of hydrolysis on gastric emptying in children. BMC Gastroenterol. 2015 Oct 15;15:137. doi: 10.1186/s12876-015-0369-0. PMID 26472544